CLINICAL TRIAL: NCT05720039
Title: A Prospective, Multicenter Randomized Controlled Trial(RCT) of the da Vinci® SP™ Surgical System vs Open Surgery in Nipple Sparing Mastectomy (NSM) Procedures
Brief Title: Robotic vs. Open NSM for Early Stage Breast Cancer
Acronym: SP NSM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISI dV SP - NSM-01
Record Dates: First submitted 2023-01-17; First posted 2023-02-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Female; Breast Cancer; Breast Cancer, Early-Onset; Breast Disease; Breast
Keywords: robotic; NSM; Nipple sparing mastectomy; da Vinci; breast cancer; mastectomy; breast; USA; robot; SP System; Single-port
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Intervention Model Description: Subjects undergo nipple-sparing mastectomy (NSM) procedures using the da Vinci SP Surgical System or open NSM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Robotic NSM with da Vinci SP (Experimental): Subjects randomized to this arm will undergo robotic NSM (RNSM) procedures
  Interventions: Device: Robotic NSM
- Open NSM (Active Comparator): Subjects randomized to this arm will undergo conventional open NSM procedures
  Interventions: Procedure: Open NSM

INTERVENTIONS:
Device: Robotic NSM — Robotic-assisted Nipple sparing mastectomy procedures
  Other Names: RNSM; SP NSM
  Arms: Robotic NSM with da Vinci SP
Procedure: Open NSM — open nipple-sparing mastectomy procedures
  Arms: Open NSM

SUMMARY:
This study evaluates the safety and effectiveness of the da Vinci SP Surgical System compared to Open NSM in Nipple Sparing Mastectomy procedures.

DETAILED DESCRIPTION:
This study is a prospective, two-arm, multi-center, randomized controlled clinical investigation between RSNM and open NSM.

This study evaluates the safety and effectiveness of the da Vinci SP Surgical System compared to Open NSM in Nipple Sparing Mastectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Female age 21 or older
* BMI < 30
* Candidate for an NSM procedure with immediate reconstruction
* Diagnosis of early stage brest cancer
* Breast ptosis ≤ Grade 2.
* Cup size ≤ C.

Exclusion Criteria:

* Previous breast surgery
* Diagnosis of metastatic breast cancer
* Prior radiation treatment to the chest
* Current smokers
* Contraindication for general anesthesia or surgery.
* Known bleeding or clotting disorder.
* Pregnant or suspected to be pregnant, or actively breastfeeding

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | Assessed during procedure
  Conversion is defined as conversion of da Vinci Xi robotic-assisted surgery to open surgery
Safety: Adverse event rates | Up to 42 days post-operatively
  Incidence of intraoperative and post-operative procedure and device-related adverse events compared to open NSM
Safety: positive surgical margin rates | Up to 42 days post-operatively
  Incidence of positive surgical margins compared to open NSM

SECONDARY OUTCOMES:
Oncological Outcomes (for cancer recurrence) | Up to 5 years
  Recurrence
Oncological Outcomes (for disease-free survival) | Up to 5 years
  Disease-free survival
Oncological Outcomes (for overall survival) | Up to 5 years
  Overall survival
Patient-Report Outcomes (BREAST-Q) | Up to 5 years
  BREAST-Q
Patient-Report Outcomes (NAC Questionnaire) | Up to 5 years
  NAC Questionnaire
Patient-Report Outcomes (EQ-5D) | Up to 1 year
  EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Gorrepati, Study Director — Intuitive
Locations (15):
- United States (15):
  - City of Hope, Irvine, California
  - Cedars-Sinai, Los Angeles, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Endeavor Health, Evanston, Illinois
  - Corewell, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Northwell Health, Lake Success, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
  - Ascension St. Columbia Mary's, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No